CLINICAL TRIAL: NCT05678543
Title: Danish Diabetes Birth Registry 2
Acronym: DDBR2
Status: Recruiting | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 1234
Record Dates: First submitted 2022-12-16; First posted 2023-01-10 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Pregnancy in Diabetic; Type 1 Diabetes; Type 2 Diabetes; Parents; Fetal Complications; Maternal Diabetes; Birth Injuries; Family
MeSH Terms: conditions — Pregnancy in Diabetics; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes, Gestational; Birth Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Months
Biospecimen Retention: Samples With DNA — Se project description
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Mothers: Pregnant women with pre existing diabetes.
- Partners: Partners to pregnant women with pre existing diabetes.
- Offspring: Offspring born to women with pre existing diabetes

SUMMARY:
Pregnancies in women with pre-existing diabetes are considered "high risk" pregnancies, poses daily clinical challenges and in terms of research - a number of unanswered questions. Therefore, the investigators wish to establish a nationwide cohort of pregnancies complicated by pre-existing diabetes - the Danish Diabetes Birth Registry (DDBR2) The DDBR2 registry comprises all types of pre-existing diabetes including T1D, T2D and other types (as MODY), generating a nationwide cohort of mother/partner/children trios with accessible registry-, clinical data and biological biobank samples. This will enable the investigators to use data longitudinally to examine short- and long-term outcomes of pregnancies in women with diabetes.

DETAILED DESCRIPTION:
During pregnancy in women with type 1 and type 2 (pre-existing) diabetes development of complications is 2-4 times higher than in the background population, as among women with pre-existing diabetes up to 50% of the offspring becomes large for gestational age (LGA), and one out of five are delivered preterm. Strict glycemic control and appropriate gestational weight gain are important for a healthy pregnancy outcome. However, a large proportion of pregnant women with diabetes do not reach the goals for glycemic control or weight gain during pregnancy.

From 1992-2000, all pregnancies in women with type 1 diabetes were reported to the Danish Diabetes Birth Registry (DDBR), which gave rise to several important international publications on perinatal outcomes and long-term follow-up studies in mother and child. During the last 20 years type 2 diabetes has become increasingly common in young women. Today up to 60% of pregnant women with pre-existing diabetes have type 2 diabetes. In Denmark we have no national surveillance of pregnancies in women with pre-existing diabetes. It is also relevant to obtain information in a national setting on partner, socioeconomic factors as well as collecting biological samples to get the information needed for a more personalized treatment of pregnant women with pre-existing diabetes.

Offspring born to women with type 1 diabetes have a higher risk of type 1 diabetes per se (5.3%) compared to the background population, but a lower risk compared to offspring of fathers with type 1 diabetes (7.8%). This fact suggests that either differences in inheritability of maternal vs. paternal susceptibility genes or maternal imprinting or maternal diabetes (i.e., the intrauterine environment) modify a child's inherited risk of developing type 1 diabetes.

For type 2 diabetes, genome-wide association studies have described approximately 250 loci being associated with type 2 diabetes. However, the genetic composition of type 2 diabetes is dominated by common alleles with small impact on the risk of disease. As opposed to type 1 diabetes, the risk of type 2 diabetes is higher in the offspring if the mother has type 2 diabetes rather than if the father has type 2 diabetes. Genetically, this can be associated with a unique parent-of-origin transmission of the risk alleles, and it relates to genetic programming during the intrauterine period.

However, the DNA sequence alone cannot explain the phenotypical variation seen in offspring born to women with diabetes. Let alone, describe how the intrauterine environment can influence the long term health of the offspring. Later in life offspring of women with diabetes faces an increased risk of obesity, pre-diabetes and type 2 diabetes, beyond what can be explained by the DNA sequence. This increase in risk of disease is for now unexplained. However, the suboptimal intrauterine environment associated with diabetes in pregnancy, may lead to epigenetic changes of the fetal DNA. Such "fetal programming of adult disease" could provide a pathogenic explanation.

Apart from genetics and epigenetics, inflammatory markers and metabolic markers of the intrauterine environment are interesting, as these have been described as altered among adolescent offspring born to women with diabetes.

Taking this into account, the possibility of predicting which offspring is at risk of later life disease is compelling and the use of proteomics, inflammatory and metabolic markers, placental markers, genetic risk scores and microRNA/small RNAs, as well as epigenetic marks, as biomarkers needs to be further explored.

Rationale for this study Pregnancies in women with pre-existing diabetes are still considered "high risk" pregnancies and pose challenges in terms of daily clinical management. Therefore, to explore this risk in a current Danish population, map the influence of both maternal and partner factors on offspring health, and comprehend how the intrauterine environment can influence both short- and long-term health of the offspring, the investigators wish to establish a nationwide cohort of pregnancies complicated by pre-existing diabetes - the Danish Diabetes Birth Registry (DDBR2).

In the DDBR2 registry the investigators wish to include data on both the woman, her partner and the child, thereby generating a nationwide cohort of mother/partner/children trios with accessible registry data, clinical data and biological samples. This will enable the investigators to use data longitudinally to examine short- and long-term outcomes of pregnancies in women with pre-existing diabetes. The DDBR2 registry will be complimented by an associated genetic, epigenetic and metabolomic interrogation seeking to illuminate possible pathogenic mechanisms that link maternal diabetes to the later life increased risk of lifestyle disease in the offspring as well as a biobank for future research.

Hypotheses of the DDBR2:

The risk of maternal and neonatal complications following a pregnancy complicated by pre-existing diabetes has decreased over the last 30 years.

Better understanding of the predictive role of socioeconomic background and maternal physical and mental health and use of technical devices prior to pregnancy can decrease the risk of an adverse pregnancy outcome.

Partner health and socioeconomic background influence pregnancy outcome. Measures of glucose from continuous glucose monitoring as predictors of adverse perinatal outcomes may be superior to HbA1c.

Epigenetic alterations in offspring cord blood reflects the intrauterine environment and can be used as markers for later life health.

Genetic risk scores for both parents and child can be used to predict risk for later life disease.

Clinical proteomics can identify novel biomarkers for maternal and offspring risk.

Micro RNA and other small RNAs can provide new insight in pathophysiology related to maternal and offspring risk.

Low-grade inflammation during pregnancy may negatively influence the glucose tolerance of the mother and perinatal outcomes.

Specific endpoints

The following endpoints apply in women with pre-existing diabetes and in their offspring in both the DDBR2 registry:

Primary endpoints Primary maternal endpoint: HbA1c levels at end of pregnancy (35 weeks) Primary offspring endpoint: Offspring birth weight adjusted for gestational age and gender (standard deviation (SD) score)

Secondary endpoints HbA1c levels during pregnancy at inclusion, 21, 33 and 35 weeks The average glucose level and percentage of time spent in the continuous glucose monitoring (CGM) target range 3.5-7.8 mmol/L, below target range (glucose <3.5 mmol/L) or above target range (glucose >7.8 mmol/L). The levels will be evaluated at night-time (24 pm to 6 am) and over 24 h, respectively, in pregnancy, during delivery and in the first one-month period after delivery.

The incidence of severe hypoglycemia in the year preceding pregnancy, during pregnancy and in the first one-month period after delivery Maternal gestational weight gain and weight retention one month after delivery In women on insulin pump therapy: insulin pump settings (mainly basal rates, carbohydrate ratio and sensitivity) in pregnancy, around delivery and the first month after delivery during lactation The prevalence of fetal overgrowth, defined as the offspring birth weight SD score >90th percentile Pregnancy complications: prevalence of induced abortion (including indication for abortion), miscarriage, gestational hypertension, preeclampsia, need for maternal corticosteroid treatment for fetal lung maturation, diabetic ketoacidosis, urinary tract infection, early preterm delivery (before 34 completed weeks), preterm delivery (before 37 completed weeks), preterm prelabour rupture of the membranes Birth complications: shoulder dystocia, birth canal trauma, mode of delivery (vaginal, cesarean section, instrumental delivery), postpartum hemorrhage, maternal death, antihypertensive treatment given one month after delivery Neonatal morbidity (neonatal hypoglycemia, jaundice, respiratory distress, transient tachypnoea, duration of stay in neonatal intensive care unit, total number of admission days), cord blood pH, stillbirths, infant death within one month Major congenital malformations (ICD10 Q00-Q99 or requiring medical or surgical treatment) Infant growth and health at one month of age Maternal and Partner Quality of Life in pregnancy and one month postpartum Maternal mental health in pregnancy and one month postpartum Average glucose level and the percentage of time in the first one-month period after delivery spent in the CGM target range 3.9-10.0 mmol/L, below target range (glucose <3.5 mmol/L) or above target range (glucose >7.8 mmol/L) at night-time (24 pm to 6 am) and over 24 h, respectively

3. Methods DDBR2 is a prospective combined clinical and register-based cohort study including all pregnant women with pre-existing diabetes aged ≥18 years in Denmark, their children and their partners corresponding to ~400 pregnant women each year (250 type 1 diabetes, 150 type 2 diabetes and 5-10 other types), a total of 2000 trios during the inclusion period. The inclusion period is from 1st Jan. 2023- 31st Dec. 2027. The registry will include data from electronic patient charts, CGM data, fetal ultra sound data, clinical data, background information on socioeconomic background, online questionnaires and biological samples.

4. Statistics A two-sided p-value <0.05 will be regarded as statistically significant in all statistical analyses.

For the primary outcomes we plan to use Mann-Whitney U test or Chi2 test. Regression analysis will be performed to determine predictors for maternal and perinatal outcomes. Sub analysis for type 1 diabetes and type 2 diabetes with and without the use of diabetes technology will be performed separately. Using a two-level approach for degree of participation, we expect a participation rate of ≈80%. In the previous DDBR registry the participation rate was 75-93% depending on inclusion site12.

5. Biological material

In the DDBR2 study the investigators wish to extract blood samples from both the parents and the offspring with the aim of answering the following research questions:

If differences in offspring cord blood methylation status is induced by intrauterine hyperglycemia, maternal obesity or hereditary predisposition.

If parental small RNAs levels during pregnancy and offspring small RNAs levels after delivery can be associated to neonatal outcome (e.g., birthweight).

If specific proteins, identified by proteomics, in either maternal, partner or offspring blood associated with maternal or neonatal morbidity.

How maternal, paternal and child genetic risk scores for type 1 diabetes, type 2 diabetes and other cardiometabolic traits (i.e., glucose levels, blood pressure, lipid levels, insulin secretion, insulin resistance, BMI, weight, waist corrected for BMI) can predict later life risk of disease.

Parent-of-origin transmission of risk alleles for type 1 and type 2 diabetes If parental and offspring levels of inflammatory cytokines, such as TNFa, IFNg, CD163, various chemokines and interleukins and vascular factors are associated with maternal or neonatal morbidity.

Parental and offspring levels of metabolic biomarkers, such as C-peptid, FGF 21, leptin, adiponectin, GDF-15, CD-59, adrenomedullin, apo-lipo protein, cortisol, cortisol binding hormone and prolactin and offspring morbidity.

Level of placental serum markers, such as PLGF, s-FLt, PAPP-A and placenta derived exosomes as predictors of pregnancy and birth outcome.

ELIGIBILITY:
Inclusion Criteria:

* Women, age ≥ 18 years
* Type 1 diabetes, type 2 diabetes or other types of pre-existing diabetes (e.g., maturity onset diabetes of the young (MODY))
* Partners of women fulfilling these inclusion criteria, age ≥ 18 years
* Offspring of women fulfilling these inclusion criteria

Exclusion Criteria:

* No proficiency in Danish or English to understand oral and written information

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: DDBR2 is a prospective combined clinical and register-based cohort study including all pregnant women with pre-existing diabetes aged ≥18 years in Denmark, their children and their partners corresponding to ~400 pregnant women each year (250 type 1 diabetes, 150 type 2 diabetes and 5-10 other types), a total of 2000 trios during the inclusion period. The inclusion period is from 1st Jan. 2023- 31st Dec. 2027. The registry will include data from electronic patient charts, CGM data, fetal ultra sound data, clinical data, background information on socioeconomic background, online questionnaires and biological samples.
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Maternal glycemic control | 35 weeks
  Maternal HbA1c (mmol/mol) levels at the end of pregnancy (35 weeks)
Offspring birthweight | 40 weeks
  Offspring birthweight (g) adjusted for gestational age and gender (standard deviation score)

CONTACTS AND LOCATIONS:
Overall Officials: Dorte M Jensen, Prof., Principal Investigator — Steno Diabetes Center Odense
Locations (4):
- Denmark (4):
  - Dept. of Obstetrics and Gynaecology, Aalborg University Hospital, Aalborg
  - Dept. of Obstetrics and Gynaecology, Aarhus Universitety Hospital, Aarhus
  - Center for Pregnant Women with Diabetes, Copenhagen University Hospital , Rigshospitalet, Copenhagen
  - Dept. of Obstetrics and Gynaecology, Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: Undecided
After the project end-date the registry data will be transferred to a future research database under the Steno Diabetes Centers. Access to this future database for external researchers is, at the moment, undecided.

REFERENCES:
- [Derived] Knorr S, Aalders J, Overgaard M, Stovring H, Mathiesen ER, Damm P, Clausen TD, Bjerre-Christensen U, Andersen LLT, Vinter C, Kofoed-Enevoldsen A, Lauenborg J, Kampmann U, Fuglsang J, Ovesen PG, Christensen TT, Sorensen A, Ringholm L, Jensen DM. Danish Diabetes Birth Registry 2: a study protocol of a national prospective cohort study to monitor outcomes of pregnancies of women with pre-existing diabetes. BMJ Open. 2024 Apr 25;14(4):e082237. doi: 10.1136/bmjopen-2023-082237. PMID 38670616